CLINICAL TRIAL: NCT04874506
Title: An Open Label Study to Assess the Safety and Clinical Efficacy of MBM-02 to Increase Survival in Patients With Newly Diagnosed Glioblastoma Multiforme (GBM)
Brief Title: MBM-02 (Tempol) for the Treatment of Glioblastoma Multiforme (GBM)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Matrix Biomed, Inc. (Industry)
Collaborators: MedStar Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MBI-10-01
Expanded Access: Available
Record Dates: First submitted 2021-05-03; First posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Glioblastoma; Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — tempol; TEMPOL-H

STUDY DESIGN:
Intervention Model Description: Three dosing regimens will be explored and represented by Cohort 1, Cohort 2, and Cohort 3.
  The first 6 patients (Cohort 1) will begin with a total daily dose (TDD) of 1000 mg of MBM-02.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Cohort 1 will receive standard of care concomitantly with1000 mg/day of MBM-02.
  Patients will receive standard of care treatment for newly diagnosed Glioblastoma multiforme consisting of four sequential periods:
  1. 1 week run-in with MBM-02 prior to radiotherapy;
  2. 6 weeks of radiotherapy and concomitant temozolomide;
  3. 4 weeks of rest post-radiotherapy and concomitant temozolomide; and
  4. Adjuvant temozolomide treatment post 4-week rest period. Patients will be administered daily MBM-02 during all four sequential periods.
  Interventions: Drug: MBM-02
- Cohort 2 (Experimental): Cohort 2 will receive standard of care concomitantly with1200 mg/day of MBM-02.
  Patients will receive standard of care treatment for newly diagnosed Glioblastoma multiforme consisting of four sequential periods:
  1. 1 week run-in with MBM-02 prior to radiotherapy;
  2. 6 weeks of radiotherapy and concomitant temozolomide;
  3. 4 weeks of rest post-radiotherapy and concomitant temozolomide; and
  4. Adjuvant temozolomide treatment post 4-week rest period. Patients will be administered daily MBM-02 during all four sequential periods.
  Interventions: Drug: MBM-02
- Cohort 3 (Experimental): Cohort 2 will receive standard of care concomitantly with1400 mg/day of MBM-02.
  Patients will receive standard of care treatment for newly diagnosed Glioblastoma multiforme consisting of four sequential periods:
  1. 1 week run-in with MBM-02 prior to radiotherapy;
  2. 6 weeks of radiotherapy and concomitant temozolomide;
  3. 4 weeks of rest post-radiotherapy and concomitant temozolomide; and
  4. Adjuvant temozolomide treatment post 4-week rest period. Patients will be administered daily MBM-02 during all four sequential periods.
  Interventions: Drug: MBM-02
- Cohort 4 (Experimental): Cohort 2 will receive standard of care concomitantly with1400 mg/day of MBM-02.
  Patients will receive standard of care treatment for newly diagnosed Glioblastoma multiforme consisting of four sequential periods:
  1. 1 week run-in with MBM-02 prior to radiotherapy;
  2. 6 weeks of radiotherapy and concomitant temozolomide;
  3. 4 weeks of rest post-radiotherapy and concomitant temozolomide; and
  4. Adjuvant temozolomide treatment post 4-week rest period. Patients will be administered daily MBM-02 during all four sequential periods.
  Interventions: Drug: MBM-02

INTERVENTIONS:
Drug: MBM-02 — Study drug will be administered orally using the capsule formulation (200 mg). The study drug will be administered 7 days a week for the entire treatment period.
  Other Names: Tempol; 4-hydroxy-tempo; 4-hydroxy-2,2,6,6-tetramethylpiperidine-1-oxyl

SUMMARY:
MBM-02 (Tempol) is an HIF-1 and HIF-2 inhibitor that is being tested as an addition to standard of care treatment that includes radiotherapy and TMZ. MBM-02's ability to increase progression free survival and decrease side effects of TMZ and radiotherapy treatment will be assessed.

DETAILED DESCRIPTION:
MBM-02 is an HIF-1 and HIF-2 inhibitor that has shown in animal models to turn back on the apoptosis process (cell death) in cancer.

Hypoxia is well documented in most solid tumors (Vaupel et al., 1991). Acute, intermittent, and cycling hypoxia are associated with inadequate blood flow, whereas chronic hypoxia is the consequence of increased oxygen diffusion distance resulting from tumor expansion (Dewhirst et al., 2008). A study by Chen and colleagues (2015) showed that cycling hypoxia and chronic hypoxia are important tumor microenvironment phenomena that limit tumor response to chemotherapy in GBM.

In hypoxic conditions observed in solid state tumors, the hypoxia inducible factors, HIF-1α and HIF-2α, are upregulated and transcribe a panel of genes associated with cancer survival and progression, such as vascular endothelial growth factor receptor (VEGFR), platelet derived growth factor (PDGF), and glucose transporter 1 (GLUT1). These factors are essential for tumor survival, thereby increasing tumor progression and decreasing apoptosis. Without the functions of the HIF family of genes, solid-state tumors could not progress and would not survive. In both Chen et al. (2015) and Sourbier et al. (2012), researchers established that the active compound in MBM-02 is an inhibitor of both HIF-1α and HIF-2α.

This is an open label multisite trial that will assess MBM-02's ability to increase progress free survival in patients receiving standard of care for glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

1. Be > 35 and ≤ 75 years of age;
2. Be newly diagnosed with glioblastoma multiforme within 4 weeks of open biopsy/resection;
3. Be histologically confirmed to have definitive GBM by partial or complete surgical resection (i.e. not by biopsy only) within 4 weeks prior to MBM-02 administration;
4. Have recovered from the effects of surgery, post-operative infection, and other complications before study registration;
5. Have a diagnostic contrast-enhanced MRI or CT scan of the brain performed preoperatively and postoperatively prior to the initiation of radiotherapy, within 28 days prior to MBM-02 administration;
6. If female and of child bearing potential, must be using an effective birth-control method as described in section 3.5;
7. If a male with a female partner of child bearing potential, adequate methods of contraception must be employed as described in section 3.5.
8. If male, no sperm donation for 90 days until after the conclusion of the study;
9. Be properly informed of the nature and risks of the clinical investigation, comply with all clinical investigation-related procedures, and sign an Informed Consent Form prior to entering the clinical investigation;
10. Be able to participate for the full term of the clinical investigation;
11. Have a Karnofsky performance status of >70;
12. Have a life expectancy ≥ 6 months; and
13. Have adequate baseline organ function (hematologic, liver, renal, nutritional and metabolic):

Hematology:

Absolute neutrophil count (ANC) ≥1.5 Hemoglobin ≥ 10 g/dL Platelets ≥ 100,000 per microliter of blood

Hepatic:

Total bilirubin ≤ 2 x ULN Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤2 x ULN

Renal:

creatinine clearance (CrCl) ≥ 60 ml/min within 2 weeks prior to registration determined by 24-hour collection or estimated by Cockcroft-Gault formula: CrCl male = [(140 - age) x (wt in kg)] [(Serum Cr mg/dl) x (72)] CrCl female = 0.85 x (CrCl male)

Exclusion Criteria:

1. Evidence of recurrent GBM or metastases detected outside of the cranial vault;
2. Patients with histone H3 K27M mutation or gliosarcoma;
3. Patients using the Optune device during study drug administration;
4. Prior cancer diagnosis other than skin basal cell or squamous cell carcinoma (non-metastatic);
5. Patients unable to undergo MRI because of non-compatible devices;
6. Oxygen dependent chronic obstructive pulmonary disease (COPD);
7. Unstable coronary artery disease (CAD);
8. Diagnosis of midline diffuse glioma (glioblastoma);
9. Insufficient biopsy tissue for full molecular profiling of the tumor;
10. Prior radiation or chemotherapy for glioblastoma or glioma;
11. Prior radiation for cancer of the head and neck that would result in an overlap of radiation fields;
12. Evidence of a significant medical illness, or a psychiatric illness/social situation that would, in the investigator's judgment, make the patient inappropriate for this study;
13. Refractory nausea and vomiting, malabsorption, biliary shunt, or significant bowel resection that would preclude adequate absorption of the study drug;
14. Have had a recent, serious, non-malignant medical complication that, in the opinion of the investigator, makes the individual unsuitable for study participation;
15. Have used an investigational drug within 28 days of the initiation of study treatment;
16. Have a history of a positive blood test for HIV;
17. At the time of screening, have a significant active medical illness which, in the opinion of the investigator, would preclude completion of the study; and
18. Body weight less than 35 kg (77 lbs.)

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | baseline to 6 months
  Clinical efficacy as measured by progression-free survival rate at six months (PFS-6). Progression-free survival will be defined as the number of days from the date of first dose to the date of earliest disease progression based on RANO criteria.

SECONDARY OUTCOMES:
Overall Survival | baseline to 24 months
  Clinical efficacy as measured by the Overall Survival (OS) rate at 12 months, 18 months, and 24 months.
Thrombocytopenia | baseline to 12 months
  Reduction in thrombocytopenia as measured by platelet count.
Neutropenia | baseline to 12 months
  Reduction in neutropenia as measured by absolute neutrophil count

OTHER OUTCOMES:
Radiation Necrosis | baseline to 3 months post-RT
  Reduction in radiation necrosis as measured by steroid dosage on the last day of RT, 1 month post-RT, and 3 months post-RT

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Watson, M.D., Principal Investigator — Georgetown University
Locations (1):
- Georgetown, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://matrixbiomed.com